CLINICAL TRIAL: NCT03376230
Title: Role of the Chemical Environment in the Pathogenesis of Inflammatory Bowel Disease
Acronym: CHIMICI
Status: Terminated | Type: Observational
Why Stopped: not enough recruitment
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2009_13; 2010-A00056-33 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Environmental risk factors; Xenobiotic detoxification
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Intestinal mucosal biopsies Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control patients
  Interventions: Other: Collect of blood, urines, and intestinal biopsies
- Crohn's disease patients
  Interventions: Other: Collect of blood, urines, and intestinal biopsies
- Ulcerative colitis patients
  Interventions: Other: Collect of blood, urines, and intestinal biopsies

INTERVENTIONS:
Other: Collect of blood, urines, and intestinal biopsies

SUMMARY:
Inflammatory Bowel Diseases (IBD) including Crohn's disease and ulcerative colitis are multifactorial diseases leading to chronic inflammation of intestinal mucosa. Their etiology is still unknown. Recently, major advances in the understanding of their pathophysiology have allowed to define them as heterogenic polygenic diseases, occurring in genetically susceptible patients. However, the whole genetic susceptibility does not explain the development of IBD and several data argue in favor of the involvement of environmental factors, which remain to be identified.

The aims of this clinical trial are:

1. As main objective: To determine the effects of environmental pollutants on intestinal homeostasis and particularly on inflammatory process and endoplasmic reticulum stress.
2. As secondary objective, to assess in human the genetic susceptibility of intestinal mucosa to environmental chemical compounds (I.e. xenobiotics), its interindividual variability, and its potential involvement in the pathogenesis of IBD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are at least 18 years old
2. Has Crohn's disease or ulcerative colitis, diagnosed, confirmed by radiological and / or endoscopic examination within 4 years or "Control" patient not suffering from inflammatory bowel disease (patient with abdominal pain and / or persistent diarrhea, or patient requiring coloscopy for cancer of the digestive tract diagnosis)
3. Patients requiring coloscopy as part of their medical follow-up
4. Social insured.

Exclusion Criteria:

1. Pregnant women
2. Breastfeeding women
3. People in emergency
4. Persons unable to understand, read and / or sign informed consent
5. Patients who recently had an intercurrent episode (eg recent diarrhea ...)
6. Persons deprived of their liberty
7. Persons protected by a legal protection status

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 600 divided into 3 groups:
  * 200 patients with ulcerative colitis
  * 200 patients with Crohn's disease
  * 200 control patients not suffering from inflammatory bowel disease and whose follow-up requires the realization of a coloscopy
Sampling Method: Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

PRIMARY OUTCOMES:
Comparison of inflammatory response of biopsies to pollutants between the 3 groups of patients. | Baseline

SECONDARY OUTCOMES:
Comparison of expression pattern of genes involved in xenobiotics detoxification in intestinal mucosa in between the 3 groups of patients. | Baseline

OTHER OUTCOMES:
Study of molecular origin and consequences of the genetic variability observed. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Desreumeaux, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU, Hôpital Claude Huriez, Lille, France

IPD SHARING:
Plan to Share IPD: Undecided